CLINICAL TRIAL: NCT03112070
Title: Post-Exercise Hypotension After Water Exercise in Older Women With Hypertension: A Randomized Crossover Clinical Trial
Brief Title: Post-Exercise Hypotension After Water Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Water Exercise
Record Dates: First submitted 2017-04-03; First posted 2017-04-13 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Postexercise Hypotension
MeSH Terms: conditions — Post-Exercise Hypotension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water aerobic exercise session (WATER) (Experimental): A continuous session of dynamic water aerobic exercise which consist of a dynamic warm-up period (5 minutes), an active exercise period (35 minutes), and a cooldown period (5 minutes) to total 45 minutes. Heart rate (HR) will be continuously measured with heart monitors (Polar) to confirm the intensity of the WATER session. The WATER intensity will be calculated according to the formula proposed by Kruel for exercise in an aquatic environment18 as follows: HR for exercise = % x (HRmax - ΔHR); % is the intensity of exercise; HRmax is the maximum HR (estimated by 220 - age); ΔHR represents the difference between resting HR on land and resting HR in the water environment. Exercise intensities: 55-60% HRmax during warm-up; 70-75% HRmax during active exercise; and 55-60% HRmax during cooldown.
  Interventions: Other: Water aerobic exercise session (WATER)
- Control session (CONTROL) (No Intervention): A 45-min session with no exercise. During this session, participants will remain seated or standing as desired. They will read, talk, and drink water, but do nothing else.

INTERVENTIONS:
Other: Water aerobic exercise session (WATER) — A continuous session of dynamic water aerobic exercise which consist of a dynamic warm-up period (5 minutes), an active exercise period (35 minutes), and a cooldown period (5 minutes) to total 45 minutes. Heart rate (HR) will be continuously measured with heart monitors (Polar) to confirm the intensity of the WATER session. The WATER intensity will be calculated according to the formula proposed by Kruel for exercise in an aquatic environment18 as follows: HR for exercise = % x (HRmax - ΔHR); % is the intensity of exercise; HRmax is the maximum HR (estimated by 220 - age); ΔHR represents the difference between resting HR on land and resting HR in the water environment. Exercise intensities: 55-60% HRmax during warm-up; 70-75% HRmax during active exercise; and 55-60% HRmax during cooldown.
  Arms: Water aerobic exercise session (WATER)

SUMMARY:
Hypertension is the most prevalent cardiovascular disease risk factor among individuals 60 years of age and older. Hypertension can be prevented and modified with lifestyle interventions that include regular exercise. Water exercise is widely recommended for older adults for a variety of health benefits, but few studies have assessed the immediate ambulatory blood pressure (BP) response to water exercise, a response termed postexercise hypotension (PEH). We will assess PEH after a session of water aerobics in physically active, older women with hypertension. Twenty-four women will be randomly assign to participate in a 45 min session of moderate intensity, water aerobics (WATER) and a 45 min land control session (CONTROL). All experimental sessions will start at 9 am sharply with 7 days between them. Subjects will left the experiments wearing an ambulatory BP monitor for the next 21 hr.

ELIGIBILITY:
Inclusion Criteria:

* resting SBP ≤ 160 mmHg and DBP ≤ 100 mmHg documented by a physician;
* 65 to 80 years of age;
* physically active on land but not water (exercising 3 or more days per week as determined by the International Physical Activity Questionnaire long-form).

Exclusion Criteria:

* any febrile condition and/or infectious diseases;
* no other chronic diseases or conditions other than hypertension;
* body mass index (BMI) > 35 kg/m2;
* active smoker;
* physical or mental limitations that prevent exercising.

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure measurements | 24-hour ambulatory blood pressure monitoring after water exercise
  BP measurements will take and monitored using a 24-hour ambulatory blood pressure monitoring (ABPM) protocol according to standard procedures. BP monitoring devices (Spacelab, Redmond, WA, USA) will be used to obtain BP over 21 hours that consiste of four measurements per hour over awake period (10 am to 10 pm) and two measurements per hour over sleep period (10 pm to 6 am). For data analysis we will calculate hourly averages for awake and sleep (during the same periods as mentioned above), and over 21 hours. SBP and DBP data are presente in two different manners: readings per hour during the day and the night periods, and the BP response determined as the difference (delta) between each hourly BP measurement from baseline after WATER compared to CONTROL.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandre Lehnen, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No